CLINICAL TRIAL: NCT00468858
Title: Phase II, Randomized, Double-blind, Placebo-controlled Study of Two Doses of WRAIR Live Attenuated Tetravalent Dengue Vaccine Formulations, Administered Six Months Apart, to Healthy Adults and Children
Brief Title: A Study of Two Doses of WRAIR Dengue Vaccine Administered Six Months Apart to Healthy Adults and Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: A-14040; WIRB number 20070071 (Other: Western Institutional Review Boards (WIRB)); 106405 (Other: GSK); T-DEN-003 (Other: MRMC/WRAIR)
Record Dates: First submitted 2007-05-01; First posted 2007-05-03 (Estimated); Results first posted 2017-06-06 (Actual); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Dengue Fever; Dengue Hemorrhagic Fever; Dengue Shock Syndrome
Keywords: Dengue; Virus; Live-attenuated; Vaccine; Dengue viral infection; Dengue Vaccine
MeSH Terms: conditions — Dengue; Severe Dengue; Virus Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- T-DEN-Post-Transfection F17 (Experimental): Post-Transfection F17, full dose
  Interventions: Biological: T-DEN-Post-Transfection F17
- T-DEN-Post-Transfection F19 (Experimental): Post-Transfection F19, full dose
  Interventions: Biological: T-DEN-Post-Transfection F19
- Placebo (Placebo Comparator): Control
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Placebo — Lyophilized, single dose vials and sterile water for
  > injection; 0.5 mL dose; Vaccination schedule: 0, 6 months
  Arms: Placebo
Biological: T-DEN-Post-Transfection F17 — Lyophilized, single dose vials and sterile water for injection; 0.5 mL dose at 0 and 6 months
  Arms: T-DEN-Post-Transfection F17
Biological: T-DEN-Post-Transfection F19 — Lyophilized, single dose vials and sterile water for injection; 0.5 mL dose at 0 and 6 months
  Arms: T-DEN-Post-Transfection F19

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of two different formulations of an investigational dengue vaccine (T-DEN) against a placebo vaccine when two doses are given six months apart to adults and children.

DETAILED DESCRIPTION:
In this study, children and adults at multiple sites in Puerto Rico will be randomly allocated to receive one of two T-DEN formulations or placebo. Subjects will be stratified by age group (a specific number of subjects in each of 4 age groups [12 months to 50 years of age] will be enrolled). The study includes 6 scheduled visits and 4 scheduled venipunctures. Safety follow-up for dengue may require unscheduled visits and venipunctures.> Multiple DEN virus serotypes are endemic in Puerto Rico and all residents are considered to be at risk for dengue. The results of this phase II study will provide a basis for identifying the vaccine formulations which elicit neutralizing antibodies to all four dengue virus serotypes in a high proportion of vaccine recipients. The most immunogenic and well tolerated candidate formulation identified in this study will be considered for advancement to phase III development.>

ELIGIBILITY:
Inclusion Criteria:>

* Subjects who the investigator believes that they and/or their parents/guardians can and will comply with the requirements of the protocol (e.g., completion of the diary cards, return for follow-up visits) should be enrolled in the study.>
* A healthy male or non-pregnant female between 12 months (mths) and 50 years (yrs) of age at the time of the first vaccination;>
* Free of obvious health problems as established by medical history and physical examination before entering into the study;>
* For children: 23mths of age, full compliance with the United States Advisory Committee on Immunization Practices (U.S. ACIP) recommended childhood immunization schedule;>
* Written informed consent obtained from the subject or a parent/guardian and assent for subjects 7-20 yrs of age;>
* If the subject is female, she must be of non-childbearing potential, i.e. either pre-menarcheal, surgically sterilized or one year post-menopausal; or, if of childbearing potential, she must be abstinent or have used adequate contraceptive precautions (i.e. intrauterine contraceptive device; condom and spermicide combination, oral contraceptives or other equivalent hormonal contraception, e.g. progestin implantable, cutaneous hormonal patch or injectable contraceptives) for 30 days (dys) prior to vaccination, have a negative pregnancy test within 48 hrs prior to vaccination and must agree to continue such precautions for 60 dys after completion of the vaccination series. Any child who begins menarche during the study period must follow the same precautions listed above, from menarche until 60 dys after the second vaccine dose.>

Exclusion Criteria:>

* Pregnant or lactating female;>
* Female planning to become pregnant or planning to discontinue abstinence or contraceptive precautions;>
* History of any neurological or behavioral disorder or seizures, with the exception of a single febrile seizure in childhood; >
* History of allergic disease/reaction likely to be exacerbated by any component of the vaccine;>
* Acute or chronic, clinically significant pulmonary, cardiovascular, hepatic, renal, hematologic or endocrine functional defect, as determined by physical examination or laboratory tests;>
* Any confirmed or suspected immunosuppressive or immunodeficient condition;>
* Acute disease at the time of enrollment (acute disease is defined as the presence of a moderate or severe illness with or without fever); note that vaccine can be administered to persons with a minor illness such as diarrhea, mild upper respiratory infection with or without low-grade febrile illness, i.e., equivalent to an oral temperature <37.5°C/<99.5°F.>
* Chronic hepatomegaly, right upper quadrant abdominal pain or tenderness;>
* Chronic splenomegaly, left upper quadrant abdominal pain or tenderness;>
* Use of any investigational or non-registered drug or vaccine other than the study vaccine within 30 dys preceding the first dose of study vaccine/placebo or planned use during the study period;>
* Planned administration of a vaccine not foreseen by the study protocol during the period starting from 30 dys before each dose of the study vaccine and ending 30 dys after; with the exception of standard infant and children "inactivated" vaccines or the inactivated influenza vaccine administered to adults or children; >
* A planned move to a location that will prohibit participating in the trial for the 12 mth duration;>
* Chronic administration (defined as more than 14 dys) of immunosuppressants or other immune-modifying drugs within 90 dys preceding the first dose or planned administration during the study period. For corticosteroids, this will mean prednisone, or equivalent, 0.5 mg/kg/day. Inhaled and topical steroids are allowed;>
* Administration of immunoglobulins and/or blood products within 90 dys preceding the first dose or planned administration during the study period;>
* Hypertension;>
* Chest pain, palpitations, dizziness, shortness of breath unrelated to asthma, arrhythmias or friction rubs;>
* Any chronic systemic drug therapy to be continued during the study period (except for vitamin/mineral supplements, routine treatment for gastro-esophageal reflux);>
* Potential adult volunteers, or parents of potential child volunteers, who do not have easy access to a fixed or mobile telephone;>
* History of chronic alcohol consumption and/or drug abuse.

Ages: 12 Months to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 636 (Actual)
Dates: Start 2007-07; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Bertran-Pasarell, MD, Principal Investigator — Dept Medicina Interna Seccion Enfermedades Infecciosas; Clemente Diaz-Perez, MD, Principal Investigator — University of PR; Ines O. Esquilin-Rivera, MD, Principal Investigator — University of PR; Evelyn Matta-Fontanet, MD, Principal Investigator — Caparra Internal Medicine Research Center; Domingo Chardon-Feliciano, MD, Principal Investigator — Ponce School of Medicine; Javier Morales-Ramirez, MD, Principal Investigator — Clinical Research PR; Luis Rodriguez-Carrasquillo, MD, Principal Investigator — Private Practice, PR; Jose Rodriguez-Santana, MD, Principal Investigator — Centro de Neumologia pediatrica; Miguel Sosa-Padilla, MD, Principal Investigator — Private Practice PR; Jose Tavarez-Valle, MD, Principal Investigator — Private Practice, PR; Alberto Santiago-Cornier, MD, Principal Investigator — Department of Molecular Medicine; Anna Quintero, MD, Principal Investigator — San Juan Batista Medical School
Locations (11):
- Puerto Rico (11):
  - San Juan Batista Medical School, Caguas
  - Private Practice, Carolina
  - St Luke's Memorial Hospital, Ponce
  - Private Practice, Rio Piedras
  - RCMI Clinical Research Center, Rio Piedras
  - Caparra Internal Medicine Research Center, Río Grande
  - Torre Medica San Vicente de Paul, San Germán
  - Clinical Research PR, San Juan
  - Centro de Neumologia Pediatricia, San Juan
  - Private Practice, San Juan
  - Dept Pediatria, Esc. De Medicina, San Juan

IPD SHARING:
Plan to Share IPD: Yes
GlaxoSmithKline

REFERENCES:
- [Derived] Bauer K, Esquilin IO, Cornier AS, Thomas SJ, Quintero Del Rio AI, Bertran-Pasarell J, Morales Ramirez JO, Diaz C, Carlo S, Eckels KH, Tournay E, Toussaint JF, De La Barrera R, Fernandez S, Lyons A, Sun W, Innis BL. A Phase II, Randomized, Safety and Immunogenicity Trial of a Re-Derived, Live-Attenuated Dengue Virus Vaccine in Healthy Children and Adults Living in Puerto Rico. Am J Trop Med Hyg. 2015 Sep;93(3):441-453. doi: 10.4269/ajtmh.14-0625. Epub 2015 Jul 14. PMID 26175027

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Control
  Placebo: Lyophilized, single dose vials and sterile water for
  > injection; 0.5 mL dose; Vaccination schedule: 0, 6 months
Period: Overall Study
Arm/Group | T-DEN-Post-Transfection F17 | T-DEN-Post-Transfection F19 | Placebo
Started | 211 | 212 | 213
Completed | 202 | 202 | 199
Not Completed | 9 | 10 | 14
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Withdrawal by Subject | 7 | 4 | 5
Not completed — Relocation | 1 | 3 | 3
Not completed — Lost to Follow-up | 1 | 2 | 5
Not completed — Other | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | T-DEN-Post-Transfection F17 | T-DEN-Post-Transfection F19 | Placebo | Total
Number analyzed (Participants) | 211 | 212 | 213 | 636
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.8 (14.10) | 12.8 (12.51) | 13.6 (13.89) | 13.4 (13.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 107 | 114 | 114 | 335
  Male | 104 | 98 | 99 | 301
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 210 | 212 | 213 | 635
  Not Hispanic or Latino | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: African heritage / African American | 2 | 1 | 2 | 5
  Race: American | 0 | 1 | 2 | 3
  Race: Dominican | 2 | 2 | 1 | 5
  Race: Hispanic | 0 | 1 | 1 | 2
  Race: Mixed | 9 | 7 | 10 | 26
  Race: Peruvian | 1 | 0 | 0 | 1
  Race: Puerto Rican | 164 | 166 | 164 | 494
  Race: White-Arabic / North African heritage | 1 | 0 | 1 | 2
  Race: White - Caucasian / European heritage | 32 | 34 | 32 | 98
Region of Enrollment [Count of Participants; unit: Participants]
  Puerto Rico | 211 | 212 | 213 | 636

OUTCOME MEASURES:

1. Primary Outcome: Safety: Incidence of All and Grade 3 Solicited Local Symptoms
Description: Incidence of all and grade 3 (prevents normal, everyday activities) solicited local and general symptoms within the 21-day follow-up period (Total vaccinated cohort)
Time Frame: Within 21 days (days 0-20) f/up period after each vaccine dose
Measure: Number; unit: number of occurances
Arm/Group | T-DEN-Post-Transfection F17 | T-DEN-Post-Transfection F19 | Placebo
Number analyzed (Participants) | 211 | 212 | 213
number of occurances
  All Grade 3 AEs | 114 | 98 | 84
  Pain - All | 55 | 60 | 48
  Pain - Grade 3 | 1 | 0 | 0
  Redness - All | 31 | 22 | 20
  Redness - Grade 3 | 6 | 2 | 5
  Swelling - All | 3 | 14 | 10
  Swelling - Grade 3 | 3 | 0 | 1
  Abdominal Pain - All | 28 | 39 | 28
  Abdominal Pain - Grade 3 | 0 | 1 | 1
  Fatigue - All | 28 | 33 | 32
  Fatigue - Grade 3 | 0 | 1 | 0
  Fever - All | 103 | 100 | 83
  Fever - Grade 3 | 10 | 13 | 9
  Headache - All | 75 | 73 | 72
  Headache - Grade 3 | 3 | 1 | 6
  Pruritus - All | 25 | 27 | 19
  Pruritus - Grade 3 | 0 | 0 | 1
  Rash - All | 18 | 20 | 10
  Rash - Grade 3 | 0 | 0 | 1
  Vomiting - All | 24 | 26 | 21
  Vomiting - Grade 3 | 0 | 1 | 1

2. Primary Outcome: Safety: Summary of Unsolicited Adverse Events Within the 31-day Post-vaccination Period
Description: Summary of unsolicited Adverse Events within the 31-day post-vaccination period by age group (total vaccinated cohort)
Time Frame: Within the 31-day (days 0-30) follow-up period after each vaccine dose
Measure: Count of Participants; unit: Participants
Arm/Group | T-DEN-Post-Transfection F17 | T-DEN-Post-Transfection F19 | Placebo
Number analyzed (Participants) | 211 | 212 | 213
Participants
  At least one symptom - age 1 - 4 years | 52 | 60 | 65
  At least one symptom - age 5 - 50 | 44 | 40 | 40
  Subject showing no unsolicited symptoms | 115 | 112 | 108

3. Primary Outcome: Safety: Occurrence of Serious Adverse Events (SAEs)
Description: Summary of SAEs, 6 months + 30 day follow-up period after last vaccine dose
Time Frame: 6 months + 30 day follow-up period after last vaccine dose
Measure: Count of Participants; unit: Participants
Arm/Group | T-DEN-Post-Transfection F17 | T-DEN-Post-Transfection F19 | Placebo
Number analyzed (Participants) | 211 | 212 | 213
Participants
  Subjects with at least 1 SAE - not related | 8 | 4 | 11
  Subject showing no SAE symptoms | 203 | 208 | 202
  Subjects with at least 1 SAE - related | 0 | 0 | 0

4. Secondary Outcome: Incidence of Suspected and Laboratory Confirmed Dengue
Description: Incidence of suspected and confirmed dengue reported during the 31-day (Days 0-30) post-vaccination period and after the 31-day period
Time Frame: 31-day (days 0-30) post-vaccination period and after 31-day period
Measure: Number; unit: dengue fever cases
Groups:
- During 31-Day Post Vaccination: F17; After 31-Day Post Vaccination Period: F17: Post-Transfection F17, full dose
  T-DEN-Post-Transfection F17: Lyophilized, single dose vials and sterile water for injection; 0.5 mL dose at 0 and 6 months
- During 31-Day Post Vaccination: F19; After 31-Day Post Vaccination Period: F19: Post-Transfection F19, full dose
  T-DEN-Post-Transfection F19: Lyophilized, single dose vials and sterile water for injection; 0.5 mL dose at 0 and 6 months
- During 31-Day Post Vaccination: Placebo; After 31-Day Post-Vaccination Period: Placebo: Control
  Placebo: Lyophilized, single dose vials and sterile water for
  > injection; 0.5 mL dose; Vaccination schedule: 0, 6 months
Arm/Group | During 31-Day Post Vaccination: F17 | During 31-Day Post Vaccination: F19 | During 31-Day Post Vaccination: Placebo | After 31-Day Post Vaccination Period: F17 | After 31-Day Post Vaccination Period: F19 | After 31-Day Post-Vaccination Period: Placebo
Number analyzed (Participants) | 211 | 212 | 213 | 211 | 212 | 213
dengue fever cases
  Dose 1: Suspected dengue fever | 3 | 3 | 0 | 3 | 3 | 3
  Dose 1: Suspected with med. attention | 3 | 3 | 0 | 3 | 3 | 3
  Dose 1: Confirmed dengue fever | 0 | 0 | 0 | 0 | 0 | 0
  Dose 2: Suspected dengue fever | 0 | 1 | 1 | 1 | 1 | 0
  Dose 2: Suspected with med. attention | 0 | 1 | 1 | 1 | 1 | 0
  Dose 2: Confirmed dengue fever | 0 | 0 | 0 | 0 | 0 | 0
  Overall Subject: Suspected dengue fever | 3 | 4 | 1 | 4 | 4 | 3
  Overall Subject: Suspected with med. attention | 3 | 4 | 1 | 4 | 4 | 3
  Overall Subject: Confirmed dengue fever | 0 | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: GMTs for Antibody Titer Above the Assay Cut Off to Each DEN Serotype for Unprimed and Primed Subjects
Description: Comparison of F17 and F19 formulations in terms of GMTs at month 7 (one month post dose 2) for each DEN type, -unprimed and primed subjects
Time Frame: at month 7 (one month post dose 2)
Measure: Mean (95% Confidence Interval); unit: titers
Arm/Group | T-DEN-Post-Transfection F17 | T-DEN-Post-Transfection F19
Number analyzed (Participants) | 211 | 212
titers
  Unprimed Subjects: DEN-1 | 130.9 [84.1 to 203.7] | 84.4 [43.6 to 163.5]
  Unprimed Subjects: DEN-2 | 218.6 [125.3 to 381.3] | 215.2 [116.7 to 396.7]
  Unprimed Subjects: DEN-3 | 124.5 [76.9 to 201.6] | 60.3 [33.0 to 110.2]
  Unprimed Subjects: DEN-4 | 377.7 [249.4 to 572.0] | 105.9 [55.8 to 201.0]
  Primed Subjects: DEN-1 | 1412.8 [1191.5 to 1675.3] | 1324.1 [1104.1 to 1587.9]
  Primed Subjects: DEN-2 | 1514.4 [1322.2 to 1734.6] | 1338.5 [1105.6 to 1620.6]
  Primed Subjects: DEN-3 | 1130.0 [920.0 to 1388.0] | 901.4 [707.6 to 1148.3]
  Primed Subjects: DEN-4 | 1228.4 [1014.1 to 1488.0] | 1020.8 [809.5 to 1287.4]

6. Secondary Outcome: Percent of Subjects With Neut. Antibody Titer Above the Assay Cut-off to All Dengue Serotypes
Description: Monovalent, bivalent, trivalent and tetravalent response for DEN neut. antibodies for unprimed and primed subjects
Time Frame: Pre-vaccination, at post dose 1, months 3 and 6 and post dose 2, month 7
Measure: Number (95% Confidence Interval); unit: % of subjects
Groups:
- F17: Pre-vaccination; F19: Pre-vaccination; Placebo: Pre-vaccination: Pre-vaccination (blood sample taken before dose 1)
- F17 PI (M3): Post-Transfection F-17 Post-dose 1, month 3
- F17 PI (M6): Post-Transfection F-17 Post-dose 1, month 6
- F17 PII (M7): Post-Transfection F-17 Post-dose 2, month 7
- F19 PI (M3): Post-Transfection F-19 Post-dose 1, month 3
- F19 PI (M6): Post-Transfection F-19 Post-dose 1, month 6
- F19 PII (M7): Post-Transfection F-19 Post-dose 2, month 7
- Placebo: PI (M3): Placebo control Post-dose 1, month 3
- Placebo: PI (M6): Placebo control Post-dose 1, month 6
- Placebo: PII (M7): Placebo control Post-dose 2, month 7
Arm/Group | F17: Pre-vaccination | F17 PI (M3) | F17 PI (M6) | F17 PII (M7) | F19: Pre-vaccination | F19 PI (M3) | F19 PI (M6) | F19 PII (M7) | Placebo: Pre-vaccination | Placebo: PI (M3) | Placebo: PI (M6) | Placebo: PII (M7)
Number analyzed (Participants) | 86 | 83 | 82 | 82 | 61 | 60 | 59 | 59 | 74 | 71 | 69 | 68
% of subjects
  Unprimed: Valence=None | 100 [95.8 to 100.0] | 53 [41.7 to 64.1] | 52.4 [41.1 to 63.6] | 2.4 [0.3 to 8.5] | 100 [94.1 to 100.0] | 50 [36.8 to 63.2] | 50.8 [37.5 to 64.1] | 5.1 [1.1 to 14.1] | 100 [95.1 to 100.0] | 95.8 [88.1 to 99.1] | 92.8 [83.9 to 97.6] | 94.1 [85.6 to 98.4]
  Unprimed: Valence=Monovalent | 0 [0 to 0] | 24.1 [15.4 to 34.7] | 23.2 [14.6 to 33.8] | 1.2 [0.0 to 6.6] | 0 [0 to 0] | 23.3 [13.4 to 36.0] | 27.1 [16.4 to 40.3] | 5.1 [1.1 to 14.1] | 0 [0 to 0] | 0 [0 to 0] | 1.4 [0.0 to 7.8] | 1.5 [0.0 to 7.9]
  Unprimed: Valence=Bivalent | 0 [0 to 0] | 4.8 [1.3 to 11.9] | 7.3 [2.7 to 15.2] | 2.4 [0.3 to 8.5] | 0 [0 to 0] | 5 [1.0 to 13.9] | 5.1 [1.1 to 14.1] | 8.5 [2.8 to 18.7] | 0 [0 to 0] | 0 [0 to 0] | 2.9 [0.4 to 10.1] | 1.5 [0.0 to 7.9]
  Unprimed: Valence=Trivalent | 0 [0 to 0] | 7.2 [2.7 to 15.1] | 7.3 [2.7 to 15.2] | 7.3 [2.7 to 15.2] | 0 [0 to 0] | 1.7 [0.0 to 8.9] | 3.4 [0.4 to 11.7] | 6.8 [1.9 to 16.5] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  Unprimed: Valence=Tetravalent | 0 [0 to 0] | 10.8 [5.1 to 19.6] | 9.8 [4.3 to 18.3] | 86.6 [77.3 to 93.1] | 0 [0 to 0] | 20 [10.8 to 32.3] | 13.6 [6.0 to 25.0] | 74.6 [61.6 to 85.0] | 0 [0 to 0] | 4.2 [0.9 to 11.9] | 2.9 [0.4 to 10.1] | 2.9 [0.4 to 10.2]
  Primed: Valence=Monovalent | 3.3 [0.7 to 9.3] | 1.1 [0.0 to 6.2] | 1.1 [0.0 to 6.2] | 0 [0 to 0] | 2.1 [0.3 to 7.5] | 0 [0 to 0] | 0 [0 to 0] | 1.1 [0.0 to 6.0] | 8.9 [4.2 to 16.2] | 3 [0.6 to 8.6] | 3 [0.6 to 8.6] | 2 [0.2 to 7.1]
  Primed: Valence=Trivalent | 1.1 [0.0 to 6.0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 2.1 [0.3 to 7.5] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 2 [0.2 to 7.1] | 1 [0.0 to 5.5]
  Primed: Valence=Bivalent | 0 [0 to 0] | 1.1 [0.0 to 6.2] | 1.1 [0.0 to 6.2] | 0 [0 to 0] | 3.2 [0.7 to 9.0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 1 [0.0 to 5.4] | 2 [0.2 to 7.1] | 0 [0 to 0] | 1 [0.0 to 5.5]
  Primed: Valence=Tetravalent | 96.5 [89.1 to 98.8] | 96.6 [90.4 to 99.3] | 97.7 [91.9 to 99.7] | 100 [95.8 to 100.0] | 92.6 [85.3 to 97.0] | 98.9 [94.2 to 100.0] | 100 [96.0 to 100.0] | 98.9 [94.0 to 100.0] | 90.1 [82.5 to 95.1] | 91.9 [84.7 to 96.4] | 89.9 [82.2 to 95.0] | 90.9 [84.4 to 95.8]
  Primed: Valence=None | 0 [0 to 0] | 1.1 [0.0 to 6.2] | 1.1 [0.0 to 6.2] | 0 [0 to 0] | 0 [0 to 0] | 1.1 [0.0 to 5.8] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 3 [0.6 to 8.6] | 5.1 [1.7 to 11.4] | 5.1 [1.7 to 11.4]

7. Secondary Outcome: Percent of Subjects With Neut. Sero-response to Each DEN Serotype
Description: Seropositivity rates for DEN neut. antibodies for unprimed and primed subjects
Time Frame: Pre-accination, at post dose 1, months 3 and 6 and post dose 2, month 7
Measure: Number (95% Confidence Interval); unit: percent of subject with attribute
Arm/Group | F17: Pre-vaccination | F17 PI (M3) | F17 PI (M6) | F17 PII (M7) | F19: Pre-vaccination | F19 PI (M3) | F19 PI (M6) | F19 PII (M7) | Placebo: Pre-vaccination | Placebo: PI (M3) | Placebo: PI (M6) | Placebo: PII (M7)
Number analyzed (Participants) | 86 | 83 | 82 | 82 | 61 | 60 | 59 | 59 | 74 | 71 | 69 | 68
percent of subject with attribute
  Unprimed: DEN-1, >10 ED50 | 0.0 [0.0 to 4.2] | 20.5 [12.4 to 30.8] | 22.0 [13.6 to 32.5] | 95.1 [88.0 to 98.7] | 0.0 [0.0 to 5.9] | 26.7 [16.1 to 39.7] | 18.6 [9.7 to 30.9] | 83.1 [71.0 to 91.6] | 0.0 [0.0 to 4.9] | 4.2 [0.9 to 11.9] | 4.3 [0.9 to 12.2] | 4.4 [0.9 to 12.4]
  Unprimed: DEN-2, >10 ED50 | 0 [0.0 to 0.0] | 26.5 [17.4 to 37.3] | 28.0 [18.7 to 39.1] | 89.0 [80.2 to 94.9] | 0.0 [0.0 to 5.9] | 43.3 [30.6 to 56.8] | 40.7 [28.1 to 54.3] | 93.2 [83.5 to 98.1] | 0.0 [0.0 to 4.9] | 4.2 [0.9 to 11.9] | 4.3 [0.9 to 12.2] | 2.9 [0.4 to 10.2]
  Unprimed: DEN-3, >10 ED50 | 0.0 [0.0 to 4.2] | 14.5 [7.7 to 23.9] | 15.9 [8.7 to 25.6] | 92.7 [84.8 to 97.3] | 0.0 [0.0 to 5.9] | 21.7 [12.1 to 34.2] | 16.9 [8.4 to 29.0] | 78.0 [65.3 to 87.7] | 0.0 [0.0 to 4.9] | 4.2 [0.9 to 11.9] | 7.2 [2.4 to 16.1] | 4.4 [0.9 to 12.4]
  Unprimed: DEN-4, >10 ED50 | 0.0 [0.0 to 4.2] | 37.3 [27.0 to 48.7] | 32.9 [22.9 to 44.2] | 97.6 [91.5 to 99.7] | 0.0 [0.0 to 5.9] | 26.7 [16.1 to 39.7] | 25.4 [15.0 to 38.4] | 86.4 [75.0 to 94.0] | 0.0 [0.0 to 4.9] | 4.2 [0.9 to 11.9] | 2.9 [0.4 to 10.1] | 4.4 [0.9 to 12.4]
  Primed: DEN-1, >10 ED50 | 97.8 [92.3 to 99.7] | 97.7 [92.0 to 99.7] | 98.9 [93.8 to 100] | 100 [95.8 to 100] | 96.8 [91.0 to 99.3] | 98.9 [94.2 to 100] | 100 [96.0 to 100] | 100 [96.0 to 100] | 94.1 [87.5 to 97.8] | 94.9 [88.6 to 98.3] | 92.9 [86.0 to 97.1] | 90.9 [83.4 to 95.8]
  Primed: DEN-2, >10 ED50 | 97.8 [92.3 to 99.7] | 96.6 [90.4 to 99.3] | 97.7 [91.9 to 99.7] | 100 [95.8 to 100] | 96.8 [91.0 to 99.3] | 98.9 [94.2 to 100] | 100 [96.0 to 100] | 98.9 [94.0 to 100] | 95.0 [88.8 to 98.4] | 93.9 [87.3 to 97.7] | 92.9 [86.0 to 97.1] | 93.9 [87.3 to 97.7]
  Primed: DEN-3, >10 ED50 | 96.7 [90.7 to 99.3] | 96.6 [90.4 to 99.3] | 97.7 [91.9 to 99.7] | 100 [95.8 to 100] | 92.6 [85.3 to 97.0] | 98.9 [94.2 to 100] | 100 [96.0 to 100] | 98.9 [94.0 to 100] | 90.1 [82.5 to 95.1] | 91.9 [84.7 to 96.4] | 90.9 [83.4 to 95.8] | 92.9 [86.0 to 97.1]
  Primed: DEN-4, >10 ED50 | 96.7 [90.7 to 99.3] | 98.9 [93.8 to 100] | 98.9 [93.8 to 100] | 100 [95.8 to 100] | 98.9 [94.2 to 100] | 98.9 [94.2 to 100] | 100 [96.0 to 100] | 98.9 [94.0 to 100] | 92.1 [85.0 to 96.5] | 93.9 [87.3 to 97.7] | 91.9 [84.7 to 96.4] | 92.9 [86.0 to 97.1]

8. Secondary Outcome: Vaccine Response to DEN Antibody at Post Dose 1, Month 3
Description: Vaccine response for DEN-1, DEN-2, DEN-3 and DEN-4 antibody
  S- = seronegative subjects (antibody titer <10 ED50 for DEN-1, 2, 3, and 4 prior to vaccination; S+ = Seropositive subjects (antibody titer >10 ED50 for DEN-1, 2, 3 and 4 prior to vaccination; Total = subjects either seropositive or seronegative at pre-vaccination
  Vaccine response defined as: For initially seronegative subjects, antibody titer >10 ED50 at PI(M3) and for initially seropositive subjects: antibody titer at PI(m3) >4 fold the pre-vaccination antibody titer
Time Frame: at month 3, post dose 1
Measure: Number (95% Confidence Interval); unit: % of subjects
Groups:
- DEN-1, F17, S-: Antibody DEN-1, Group F17, Pre-vaccination status = S-
- DEN-1, F17, S+: Antibody DEN-1, Group F17, Pre-vaccination status = S+
- DEN-1, F17, Total: Antibody DEN-1, Group F17, Pre-vaccination status = Total
- DEN-1, F19, S-: Antibody DEN-1, Group F19, Pre-vaccination status = S-
- DEN-1, F19, S+: Antibody DEN-1, Group F19, Pre-vaccination group = S+
- DEN-1, F19, Total: Antibody DEN-1, Group F19, Pre-vaccination status = Total
- DEN-1, Placebo, S-: Antibody DEN-1, Placebo group, Pre-vaccination status = S-
- DEN-1, Placebo, S+: Antibody DEN-1, Placebo group, Pre-vaccination status = S+
- DEN-1, Placebo, Total: Antibody DEN-1, Placebo group, Pre-vaccination status = Total
- DEN-2, F17, S-: Antibody DEN-2, Group F17, Pre-vaccination status = S-
- DEN-2, F17, S+: Antibody DEN-2, Group F17, Pre-vaccination status = S+
- DEN-2, F17, Total: Antibody DEN-2,. Group F17, Pre-vaccination status = Total
- DEN-2, F19, S-: Antibody DEN-2, Group F19, Pre-vaccination status = S-
- DEN-2, F19, S+: Antibody DEN-2, Group F19, Pre-vaccination status = S+
- DEN-2, F19, Total: Antibody DEN-2, Group F19, Pre-vaccination status = Total
- DEN-2, Placebo, S-: Antibody DEN-2, Placebo group, Pre-vaccination status = S-
- DEN-2, Placebo, S+: Antibody DEN-2, Placebo group, Pre-vaccination status = S+
- DEN-2, Placebo, Total: Antibody DEN-2, Placebo group, Pre-vaccination status = Total
- DEN-3, F17, S-: Antibody DEN-3, Group F17, Pre-vaccination status = S-
- DEN-3, F17, S+: Antibody DEN-3, Group F17, Pre-vaccination status = S+
- DEN-3, F17, Total: Antibody DEN-3, Group F17, Pre-vaccination status = Total
- DEN-3, F19, S-: Antibody DEN-3, Group F19, Pre-vaccination status = S-
- DEN-3, F19, S+: Antibody DEN-3, Group F19, Pre-vaccination status = S+
- DEN-3, F19, Total: Antibody DEN-3, Group F19, Pre-vaccination status = Total
- DEN-3, Placebo, S-: Antibody DEN-3, Placebo group, Pre-vaccination status = S-
- DEN-3, Placebo, S+: Antibody DEN-3, Placebo group, Pre-vaccination status = S+
- DEN-3, Placebo, Total: Antibody DEN-3, Placebo group, Pre-vaccination status = Total
- DEN-4, F17, S-: Antibody DEN-4, Group F17, Pre-vaccination status = S-
- DEN-4, F17, S+: Antibody DEN-4, Group F17, Pre-vaccination status = S+
- DEN-4, F17, Total: Antibody DEN-4, Group F17, Pre-vaccination status = Total
- DEN-4, F19, S-: Antibody DEN-4, Group F19, Pre-vaccination status = S-
- DEN-4, F19, S+: Antibody DEN-4, Group F19, Pre-vaccination status = S+
- DEN-4, F19, Total: Antibody DEN-4, Group F19, Pre-vaccination status = Total
- DEN-4, Placebo, S-: Antibody DEN-4, Placebo group, Pre-vaccination status = S-
- DEN-4, Placebo, S+: Antibody DEN-4, Placebo group, Pre-vaccination status = S+
- DEN-4, Placebo, Total: Antibody DEN-4, Placebo group, Pre-vaccination status = Total
Arm/Group | DEN-1, F17, S- | DEN-1, F17, S+ | DEN-1, F17, Total | DEN-1, F19, S- | DEN-1, F19, S+ | DEN-1, F19, Total | DEN-1, Placebo, S- | DEN-1, Placebo, S+ | DEN-1, Placebo, Total | DEN-2, F17, S- | DEN-2, F17, S+ | DEN-2, F17, Total | DEN-2, F19, S- | DEN-2, F19, S+ | DEN-2, F19, Total | DEN-2, Placebo, S- | DEN-2, Placebo, S+ | DEN-2, Placebo, Total | DEN-3, F17, S- | DEN-3, F17, S+ | DEN-3, F17, Total | DEN-3, F19, S- | DEN-3, F19, S+ | DEN-3, F19, Total | DEN-3, Placebo, S- | DEN-3, Placebo, S+ | DEN-3, Placebo, Total | DEN-4, F17, S- | DEN-4, F17, S+ | DEN-4, F17, Total | DEN-4, F19, S- | DEN-4, F19, S+ | DEN-4, F19, Total | DEN-4, Placebo, S- | DEN-4, Placebo, S+ | DEN-4, Placebo, Total
Number analyzed (Participants) | 84 | 37 | 121 | 63 | 38 | 101 | 77 | 43 | 120 | 85 | 33 | 118 | 63 | 45 | 108 | 76 | 43 | 119 | 85 | 36 | 121 | 66 | 45 | 111 | 81 | 39 | 120 | 85 | 42 | 127 | 61 | 49 | 110 | 79 | 45 | 124
% of subjects | 20.2 [12.3 to 30.4] | 54.1 [36.9 to 70.5] | 30.6 [22.5 to 39.6] | 30.2 [19.2 to 43.0] | 73.7 [56.9 to 86.6] | 46.5 [36.5 to 56.7] | 7.8 [2.9 to 16.2] | 7.0 [1.5 to 19.1] | 7.5 [3.5 to 13.8] | 25.9 [17.0 to 36.5] | 63.6 [45.1 to 79.6] | 36.4 [27.8 to 45.8] | 46.0 [33.4 to 59.1] | 64.4 [48.8 to 78.1] | 53.7 [43.8 to 63.3] | 3.9 [0.8 to 11.1] | 14.0 [5.3 to 27.9] | 7.6 [3.5 to 13.9] | 15.3 [8.4 to 24.7] | 61.1 [43.5 to 76.9] | 28.9 [21.0 to 37.9] | 28.8 [18.3 to 41.3] | 62.2 [46.5 to 76.2] | 42.3 [33.0 to 52.1] | 6.2 [2.0 to 13.8] | 5.1 [0.6 to 17.3] | 5.8 [2.4 to 11.6] | 38.8 [28.4 to 50.0] | 52.4 [36.4 to 68.0] | 43.3 [34.5 to 52.4] | 27.9 [17.1 to 40.8] | 65.3 [50.4 to 78.3] | 44.5 [35.1 to 54.3] | 7.6 [2.8 to 15.8] | 11.1 [3.7 to 24.1] | 8.9 [4.5 to 15.3]

9. Secondary Outcome: Vaccine Response to DEN Antibody at Post Dose 2, Month 7
Description: Vaccine response for DEN-1, DEN2, DEN-3, DEN-4 antibody at post dose 2, month 7
Time Frame: at month 7, post dose 2
Measure: Number (95% Confidence Interval); unit: % of subjects
Arm/Group | DEN-1, F17, S- | DEN-1, F17, S+ | DEN-1, F17, Total | DEN-1, F19, S- | DEN-1, F19, S+ | DEN-1, F19, Total | DEN-1, Placebo, S- | DEN-1, Placebo, S+ | DEN-1, Placebo, Total | DEN-2, F17, S- | DEN-2, F17, S+ | DEN-2, F17, Total | DEN-2, F19, S- | DEN-2, F19, S+ | DEN-2, F19, Total | DEN-2, Placebo, S- | DEN-2, Placebo, S+ | DEN-2, Placebo, Total | DEN-3, F17, S- | DEN-3, F17, S+ | DEN-3, F17, Total | DEN-3, F19, S- | DEN-3, F19, S+ | DEN-3, F19, Total | DEN-3, Placebo, S- | DEN-3, Placebo, S+ | DEN-3, Placebo, Total | DEN-4, F17, S- | DEN-4, F17, S+ | DEN-4, F17, Total | DEN-4, F19, S- | DEN-4, F19, S+ | DEN-4, F19, Total | DEN-4, Placebo, S- | DEN-4, Placebo, S+ | DEN-4, Placebo, Total
Number analyzed (Participants) | 83 | 35 | 118 | 61 | 37 | 98 | 74 | 43 | 117 | 84 | 32 | 116 | 62 | 42 | 104 | 73 | 43 | 116 | 84 | 34 | 118 | 64 | 43 | 107 | 78 | 39 | 117 | 84 | 40 | 124 | 60 | 48 | 108 | 76 | 45 | 121
% of subjects | 95.2 [88.1 to 98.7] | 60.0 [42.1 to 76.1] | 84.7 [77.0 to 90.7] | 83.6 [71.9 to 91.8] | 75.7 [58.8 to 88.2] | 80.6 [71.4 to 87.9] | 6.8 [2.2 to 15.1] | 11.6 [3.9 to 25.1] | 8.5 [4.2 to 15.2] | 89.3 [80.6 to 95.0] | 71.9 [53.3 to 86.3] | 84.5 [76.6 to 90.5] | 93.5 [84.3 to 98.2] | 64.3 [48.0 to 78.4] | 81.7 [72.9 to 88.6] | 4.1 [0.9 to 11.5] | 14.0 [5.3 to 27.9] | 7.8 [3.6 to 14.2] | 92.9 [85.1 to 97.3] | 47.1 [29.8 to 64.9] | 79.7 [71.3 to 86.5] | 79.7 [67.8 to 88.7] | 48.8 [33.3 to 64.5] | 67.3 [57.5 to 76.0] | 9.0 [3.7 to 17.6] | 15.4 [5.9 to 30.5] | 11.1 [6.1 to 18.3] | 97.6 [91.7 to 99.7] | 57.5 [40.9 to 73.0] | 84.7 [77.1 to 90.5] | 86.7 [75.4 to 94.1] | 68.8 [53.7 to 81.3] | 78.7 [69.8 to 86.0] | 7.9 [3.0 to 16.4] | 6.7 [1.4 to 18.3] | 7.4 [3.5 to 13.7]

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | T-DEN-Post-Transfection F17 | T-DEN-Post-Transfection F19 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/211 | 0/212 | 0/213
Serious Adverse Events (participants affected / at risk) | 8/211 | 4/212 | 11/213
Other Adverse Events (participants affected / at risk) | 90/211 | 93/212 | 93/213
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | T-DEN-Post-Transfection F17 (N=211) | T-DEN-Post-Transfection F19 (N=212) | Placebo (N=213)
Cellulitis (face) (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cellulitis orbital (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Dengue fever (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Acute gastroenteritis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Acute viral gastroenteritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Tonsillitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Presumptive viral syndrome (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Acute bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Bronchial asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Ureteral calculus (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | T-DEN-Post-Transfection F17 (N=211) | T-DEN-Post-Transfection F19 (N=212) | Placebo (N=213)
Pain (General disorders) | 25 (25) | 34 (34) | 31 (31) — Dose 1
Redness (Skin and subcutaneous tissue disorders) | 15 (15) | 15 (15) | 12 (12) — Dose 1
Swelling (General disorders) | 8 (8) | 7 (7) | 6 (6) — Dose 1
Pain (General disorders) | 30 (30) | 26 (26) | 17 (17) — Dose 2
Redness (Skin and subcutaneous tissue disorders) | 16 (16) | 7 (7) | 8 (8) — Dose 2
Swelling (Metabolism and nutrition disorders) | 10 (10) | 7 (7) | 4 (4) — Dose 2
Abdominal pain (Gastrointestinal disorders) | 18 (18) | 26 (26) | 17 (17) — Dose 1
Fatigue (General disorders) | 17 (17) | 26 (26) | 18 (18) — Dose 1
Fever (axillary) (General disorders) | 52 (52) | 54 (54) | 47 (47) — Dose 1
Headache (Nervous system disorders) | 41 (41) | 49 (49) | 45 (45) — Dose 1
Pruritus (Skin and subcutaneous tissue disorders) | 20 (20) | 19 (19) | 13 (13) — Dose 1
Rash (Skin and subcutaneous tissue disorders) | 13 (13) | 16 (16) | 9 (9) — Dose 1
Vomiting (Gastrointestinal disorders) | 13 (13) | 15 (15) | 14 (14) — Dose 1
Abdominal pain (Gastrointestinal disorders) | 10 (10) | 13 (13) | 11 (11) — Dose 2
Fatigue (General disorders) | 11 (11) | 7 (7) | 14 (14) — Dose 2
Fever (axillary) (General disorders) | 51 (51) | 46 (46) | 36 (36) — Dose 2
Headache (Nervous system disorders) | 34 (34) | 24 (24) | 27 (27) — Dose 2
Pruritus (Skin and subcutaneous tissue disorders) | 5 (5) | 8 (8) | 6 (6) — Dose 2
Rash (Skin and subcutaneous tissue disorders) | 5 (5) | 4 (4) | 1 (1) — Dose 2
Vomiting (Gastrointestinal disorders) | 11 (11) | 11 (11) | 7 (7) — Dose 2
Ear congestion (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) — Ages 1 to 4
Ear pain (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 2 (2) — Ages 1 to 4
Conjunctivitis (Infections and infestations) | 2 (2) | 4 (4) | 2 (2) — Ages 1 to 4
Photophobia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) — Ages 1 to 4
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) — Ages 1 to 4
Abdominal pain (upper) (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) — Ages 1 to 4
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) — Ages 1 to 4
Diarrhea (Gastrointestinal disorders) | 8 (8) | 6 (6) | 5 (5) — Ages 1 to 4
Enteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) — Ages 1 to 4
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1) — Ages 1 to 4
Injection site reaction (General disorders) | 1 (1) | 0 (0) | 0 (0) — Ages 1 to 4
Irritability (General disorders) | 0 (0) | 1 (1) | 0 (0) — Ages 1 to 4
Pyrexia (General disorders) | 2 (2) | 4 (4) | 1 (1) — Ages 1 to 4
Thirst (General disorders) | 0 (0) | 0 (0) | 1 (1) — Ages 1 to 4
Food allergy (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) — Ages 1 to 4
Abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) — Ages 1 to 4
Bronchiolitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) — Ages 1 to 4
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) — Ages 1 to 4
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) — Ages 1 to 4
Croup infectious (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) — Ages 1 to 4
Ear infection (Infections and infestations) | 0 (0) | 2 (2) | 2 (2) — Ages 1 to 4
Gastroenteritis (Gastrointestinal disorders) | 2 (2) | 2 (2) | 3 (3) — Ages 1 to 4
Gastroenteritis viral (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) — Ages 1 to 4
Genital candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) — Ages 1 to 4
Impetigo (Infections and infestations) | 1 (1) | 4 (4) | 3 (3) — Ages 1 to 4
Infected bites (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) — Ages 1 to 4
Infection parasitic (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) — Ages 1 to 4
Nasopharyngitis (Infections and infestations) | 13 (13) | 6 (6) | 16 (16) — Ages 1 to 4
Otitis externa (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) — Ages 1 to 4
Otitis media (Infections and infestations) | 3 (3) | 3 (3) | 4 (4) — Ages 1 to 4
Otitis media acute (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) — Ages 1 to 4
Parasitic gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) — Ages 1 to 4
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) — Ages 1 to 4
Pneumonia (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) — Ages 1 to 4
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) — Ages 1 to 4
Sinusitis (Infections and infestations) | 1 (1) | 4 (4) | 2 (2) — Ages 1 to 4
Subcutaneous abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) — Ages 1 to 4
Tonsillitis (Infections and infestations) | 1 (1) | 2 (2) | 1 (1) — Ages 1 to 4
Upper respiratory tract infection (Infections and infestations) | 12 (12) | 21 (21) | 21 (21) — Ages 1 to 4
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) — Ages 1 to 4
Viral infection (Infections and infestations) | 3 (3) | 1 (1) | 2 (2) — Ages 1 to 4
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) — Ages 1 to 4
Bruns first degree (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) — Ages 1 to 4
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) — Ages 1 to 4
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) — Ages 1 to 4
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) — Ages 1 to 4
Scratch (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) — Ages 1 to 4
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) — Ages 1 to 4
Tooth injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) — Ages 1 to 4
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) — Ages 1 to 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) — Ages 1 to 4
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) — Ages 1 to 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) — Ages 1 to 4
Crying (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) — Ages 1 to 4
Psychomotor hyperactivity (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) — Ages 1 to 4
Aggression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) — Ages 1 to 4
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) — Ages 1 to 4
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 4 (4) — Ages 1 to 4
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 0 (0) — Ages 1 to 4
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 8 (8) | 5 (5) — Ages 1 to 4
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3) | 4 (4) — Ages 1 to 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2) — Ages 1 to 4
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) — Ages 1 to 4
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 1 (1) — Ages 1 to 4
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) — Ages 1 to 4
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) — Ages 1 to 4
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (2) — Ages 1 to 4
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) — Ages 1 to 4
Rash generalized (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) — Ages 1 to 4
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) — Ages 1 to 4
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) — Ages 1 to 4
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) — Ages 1 to 4
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) — Ages 5 - 50
Conuunctivitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) — Ages 5 - 50
Conjunctivitis allergic (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) — Ages 5 - 50
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 1 (1) — Ages 5 - 50
Ocular hyperaemia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) — Ages 5 - 50
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) — Ages 5 - 50
Anal pruritus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) — Ages 5 - 50
Diarrhea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (2) — Ages 5 - 50
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) — Ages 5 - 50
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) — Ages 5 - 50
Gastritis (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) — Ages 5 - 50
Gastroesophageal reflux desease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) — Ages 5 - 50
Sensitivity of teeth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) — Ages 5 - 50
Tooth development disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) — Ages 5 - 50
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) — Ages 5 - 50
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0) — Ages 5 - 50
Exercise tolerance decreased (General disorders) | 1 (1) | 0 (0) | 0 (0) — Ages 5 - 50
Influenza like symptoms (General disorders) | 0 (0) | 0 (0) | 1 (1) — Ages 5 - 50
Injection site haematoma (General disorders) | 0 (0) | 0 (0) | 1 (1) — Ages 5 - 50
Injection site pruritus (General disorders) | 0 (0) | 0 (0) | 1 (1) — Ages 5 - 50
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) — Ages 5 - 50
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) — Ages 5 - 50
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) — Ages 5 - 50
Seasonal allergy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) — Ages 5 - 50
Abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) — Ages 5 - 50
Acute sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) — Ages 5 - 50
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) — Ages 5 - 50
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) — Ages 5 - 50
Enterobiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) — Ages 5 - 50
Fungal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) — Ages 5 - 50
Gastroenteritis (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) — Ages 5 - 50
Gastroenteritis viral (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) — Ages 5 - 50
Gingival abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) — Ages 5 - 50
Impetigo (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) — Ages 5 - 50
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) — Ages 5 - 50
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) — Ages 5 - 50
Otitis media (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) — Ages 5 - 50
Pharyngitis (Infections and infestations) | 3 (3) | 3 (3) | 5 (5) — Ages 5 - 50
Rhinitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) — Ages 5 - 50
Sinusitis (Infections and infestations) | 1 (1) | 2 (2) | 3 (3) — Ages 5 - 50
Tinea versicolour (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) — Ages 5 - 50
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) — Ages 5 - 50
Upper respiratory tract infection (Infections and infestations) | 7 (7) | 8 (8) | 7 (7) — Ages 5 - 50
Viral infection (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) — Ages 5 - 50
Viral pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) — Ages 5 - 50
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) — Ages 5 - 50
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) — Ages 5 - 50
Joint sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) — Ages 5 - 50
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (3) | 1 (1) — Ages 5 - 50
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) — Ages 5 - 50
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) — Ages 5 - 50
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) — Ages 5 - 50
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 4 (4) — Ages 5 - 50
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) — Ages 5 - 50
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) — Ages 5 - 50
Dysgeusia (Nervous system disorders) | 2 (2) | 1 (1) | 3 (3) — Ages 5 - 50
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2) — Ages 5 - 50
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) — Ages 5 - 50
Psychomotor hyperactivity (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) — Ages 5 - 50
Insomnia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) — Ages 5 - 50
Bladder pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) — Ages 5 - 50
Breast tenderness (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) — Ages 5 - 50
Ovarian disorder (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) — Ages 5 - 50
Penis disorder (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) — Ages 5 - 50
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) — Ages 5 - 50
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 1 (1) — Ages 5 - 50
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2) — Ages 5 - 50
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2) | 0 (0) — Ages 5 - 50
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (4) | 2 (2) — Ages 5 - 50
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2) | 2 (2) — Ages 5 - 50
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) — Ages 5 - 50
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 3 (3) — Ages 5 - 50
Dermititis allergic (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) — Ages 5 - 50
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) — Ages 5 - 50
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) — Ages 5 - 50
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) — Ages 5 - 50
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) — Ages 5 - 50
Rash papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) — Ages 5 - 50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No